CLINICAL TRIAL: NCT04390672
Title: A Randomized Controlled Trial to Compare the Safety and Efficacy of siroliMUs-eLuTIng Biodegradable Polymer ulTrA-thin Stent (SUPRAFLEX Cruz) and Everolimus-eLuting Biodegradable Polymer Stent (SYNERGY) in treatmENT for Three-vessel Coronary Artery Disease: Multivessel TALENT
Brief Title: Multivessel TALENT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Patrick Serruys, Established Professor of Interventional Medicine and Innovation, National University of Ireland, Galway (NUIG), Galway, Ireland, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUIG-2020-002
Record Dates: First submitted 2020-05-01; First posted 2020-05-15 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arterial Occlusive Diseases; Vascular Diseases
Keywords: multi-vessel coronary artery disease; revascularization; quantitative flow ratio; fractional flow reserve; instant wave-free ratio; SYNTAX score; prasugrel monotherapy; ultra-thin strut sirolimus-eluting coronary stent
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUPRAFLEX Cruz (Experimental): Percutaneous Coronary Intervention with the SUPRAFLEX Cruz Sirolimus Eluting Bioabsorbable Polymer Coronary Stent System. It is a balloon expandable sirolimus eluting stent with an bioabsorbable polymer coating.
  Interventions: Device: SUPRAFLEX Cruz
- SYNERGY (Active Comparator): Percutaneous Coronary Intervention with the SYNERGY EES (Everolimus Eluting) Coronary Stent System. The stents are balloon expandable drug eluting stents using everolimus with an bioabsorbable polymer coating.
  Interventions: Device: SYNERGY

INTERVENTIONS:
Device: SUPRAFLEX Cruz — Percutaneous Coronary Intervention for multivessel disease
  Arms: SUPRAFLEX Cruz
Device: SYNERGY — Percutaneous Coronary Intervention for multivessel disease
  Arms: SYNERGY

SUMMARY:
Multivessel TALENT is a prospective, randomized, multi-center study comparing clinical outcomes between SUPRAFLEX Cruz and SYNERGY in approximately 1550 patients with de-novo three vessel disease undergoing percutaneous coronary intervention (PCI). Patients will be treated according to "state of art PCI"; not only treatment strategies based on the latest ESC guideline, such as SYNTAX Score II recommendation, Heart Team discussion, post-procedure intravascular imaging optimization, cholesterol reduction by statin or PCSK-9 inhibitor, but also exploratory treatment strategies based on the latest evidence, such as physiological assessment using quantitative flow ratio and prasugrel monotherapy following 1-month dual antiplatelet therapy after PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients' ≥18 years.
2. At least 1 stenosis (angiographic, visually determined de novo lesions with ≥50% DS) in all 3 major epicardial territories (LAD and/or side branch, LCX and/or side branch, RCA and/or side branch) supplying viable myocardium without left main involvement.
3. The vessel should have a reference vessel diameter ranging from ≥2.25 mm to ≤4.50 mm (no limitation on the number of treated lesions, vessels, or lesion length).
4. Patients with chronic coronary syndrome or stabilized acute coronary syndromes.
5. All anatomical SYNTAX Scores are eligible for initial screening with the SYNTAX Score II, provided that the SYNTAX Score II recommends equipoise risk (PCI or CABG) or PCI only.
6. Patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Ethical Committee and is willing to comply with all protocol-required evaluations.
7. Agree with conditional longer follow up from 2 to 5 years with one phone contact yearly.

Exclusion Criteria:

1. Under the age of 18.
2. Unable to give informed consent.
3. Patient is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential according to local practice).
4. Known contraindication to medications such as Aspirin, Heparin, Bivalirudin, Prasugrel and Ticagrelor.
5. Prior PCI or prior CABG.
6. Ongoing ST-elevation myocardial infarction (STEMI).
7. Cardiogenic shock is also an exclusion criteria.
8. Concurrent medical condition with a life expectancy of less than 2 years.
9. Currently participating in another trial and not yet at its primary endpoint.
10. Patient with both ostial LAD and ostial LCX stenosis, or left main stenosis.
11. Previous intracranial haemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1550 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a composite of all cause death, any stroke, any myocardial infarction (MI), and any (repeat) revascularisation | 12 months post-procedure
  a non-inferiority comparison of Patient-oriented Composite Endpoint (POCE) of the SUPRAFLEX Cruz cohort to the SYNERGY cohort at 12 months post-procedure. POCE is a composite clinical endpoint of:
  * All cause death;
  * Any stroke, Modified Rankin Scale (MRS ≥1);
  * Any myocardial infarction (MI);
  * Any (repeat) revascularisation

SECONDARY OUTCOMES:
Number of vessels with a composite of vessel-related cardiovascular death, vessel-related MI, or CPI-TVR (clinically and physiologically-indicated-Target vessel revascularisation) | 24 months post-procedure
  a superiority comparison in the as treated population (per vessel level) of the vessel-oriented composite endpoints (VOCE).
  VOCE is a composite clinical endpoint of:
  * Vessel-related cardiovascular death;
  * Vessel-related MI;
  * CPI-TVR (clinically and physiologically-indicated-Target vessel revascularisation).
Number of participants with a composite of all cause death, any stroke, any myocardial infarction (MI), and any (repeat) revascularisation | 24 months post-procedure
  a comparison of Patient-oriented Composite Endpoint (POCE) of the SUPRAFLEX Cruz cohort to the SYNERGY cohort at 24 months post-procedure. POCE is a composite clinical endpoint of:
  * All cause death;
  * Any stroke, Modified Rankin Scale (MRS ≥1);
  * Any myocardial infarction (MI);
  * Any (repeat) revascularisation
Number of participants with all cause death | 12 and 24 months post-procedure
  a comparison of numbers of participants with all cause death
Number of Participants with any stroke | 12 and 24 months post-procedure
  a comparison of numbers of participants with any stroke
Number of Participants with any myocardial infarction | 12 and 24 months post-procedure
  a comparison of numbers of participants with any myocardial infarction
Number of Participants with any (repeat) revascularisation | 12 and 24 months post-procedure
  a comparison of number of participants with any (repeat) revascularisation
Number of vessels with vessel-related cardiovascular death | 12 and 24 months post-procedure
  a comparison of numbers of vessels with vessel-related cardiovascular death
Number of vessels with vessel-related MI | 12 and 24 months post-procedure
  a comparison of numbers of vessels with vessel-related MI
Number of vessels with CPI-TVR (clinically and physiologically-indicated-Target vessel revascularisation) | 12 and 24 months post-procedure
  a comparison of numbers of vessels with CPI-TVR (clinically and physiologically-indicated-Target vessel revascularisation)
Number of participants with a composite of cardiovascular death, target vessel MI and clinically-indicated target lesion revascularization | 12 and 24 months post-procedure
  a comparison of numbers of participants with TLF / DOCE defined as cardiovascular death, target vessel MI and clinically-indicated target lesion revascularisation
Number of participants with a composite of cardiovascular death, target vessel MI and clinically-indicated target vessel revascularisation | 12 and 24 months post-procedure
  a comparison of numbers of participants with TVF defined as cardiovascular death, target vessel MI and clinically-indicated target vessel revascularisation
Number of participants with cardiovascular death | 12 and 24 months post-procedure
  a comparison of numbers of participants with cardiovascular death
Number of participants with target vessel MI | 12 and 24 months post-procedure
  a comparison of numbers of participants with target vessel MI
Number of participants with clinically-indicated target lesion revascularisation | 12 and 24 months post-procedure
  a comparison of numbers of participants with clinically-indicated target lesion revascularisation
Number of participants with Definite/Probable Stent thrombosis | 12 and 24 months post-procedure
  a comparison of numbers of participants with Definite/Probable Stent thrombosis
Number of participants with device success | 7days post-procedure
  a comparison of numbers of participants with device success
Number of participants with procedure success | 7days post-procedure
  a comparison of numbers of participants with procedure success (Device success + free from POCE at discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W. Serruys, MD, PhD, Study Chair — National University of Ireland, Galway; William Wijns, MD, PhD, Study Chair — National University of Ireland, Galway; Yoshinobu Onuma, MD, PhD, Study Chair — National University of Ireland, Galway; Helge Moellmann, MD, Principal Investigator — St. Johannes Hospital; Manel Sabate, MD, PhD, Principal Investigator — Hospital Clínic of Barcelona; Azfar Zaman, MD, Principal Investigator — Freeman Hospital and Newcastle University
Locations (1):
- NUIG, Galway, Ireland

REFERENCES:
- [Derived] Kageyama S, Revaiah PC, Tsung-Ying T, Miyashita K, Tobe A, O'Leary N, Reiber JHC, Tu S, Zaman A, Sabate M, Mollmann H, Sharif F, Lemoine J, Wlodarczak A, Garg S, Onuma Y, Serruys PW. Diffuseness of coronary artery disease impacts on immediate hemodynamic and predicted clinical outcomes. Sci Rep. 2025 Jan 17;15(1):2228. doi: 10.1038/s41598-025-85872-9. PMID 39825017
- [Derived] Ninomiya K, Serruys PW, Garg S, Hara H, Masuda S, Kageyama S, Kotoku N, Sevestre E, Kumar A, O'Kane P, Zaman A, Farah B, Magro M, Oemrawsingh RM, Mollmann H, Meneveau N, Achenbach S, Lemoine J, Allali A, Gallagher S, Wykrzykowska J, Lesiak M, Silvestri M, Wijns W, Sharif F, Onuma Y. The Utility of the SYNTAX Score II and SYNTAX Score 2020 for Identifying Patients with Three-Vessel Disease Eligible for Percutaneous Coronary Intervention in the Multivessel TALENT Trial: A Prospective Pilot Experience. Rev Cardiovasc Med. 2022 Apr 8;23(4):133. doi: 10.31083/j.rcm2304133. eCollection 2022 Apr. PMID 39076220
- [Derived] Hara H, Gao C, Kogame N, Ono M, Kawashima H, Wang R, Morel MA, O'Leary N, Sharif F, Mollmann H, Reiber JHC, Sabate M, Zaman A, Wijns W, Onuma Y, Serruys PW. A randomised controlled trial of the sirolimus-eluting biodegradable polymer ultra-thin Supraflex stent versus the everolimus-eluting biodegradable polymer SYNERGY stent for three-vessel coronary artery disease: rationale and design of the Multivessel TALENT trial. EuroIntervention. 2020 Dec 18;16(12):e997-e1004. doi: 10.4244/EIJ-D-20-00772. PMID 32928717